CLINICAL TRIAL: NCT02537860
Title: Paravertebral Block for Inguinal Hernia Repair in Elderly: Randomized Double-blinded Clinical Trial
Brief Title: Paravertebral Block for Inguinal Hernia Repair in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Chairperson of Anesthesia and Pain Management Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08252015
Record Dates: First submitted 2015-08-25; First posted 2015-09-02 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Inguinal Hernia Repair
MeSH Terms: interventions — inulin trinicotinate monomethochloride; Herniorrhaphy; Fentanyl; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Three PVB injections (Experimental): Patients will receive three PVB injections from T12 to L2 and placebo at T11 and L3
  Interventions: Other: Paravertebral block injections from T12 to L2; Other: Placebo at T11 and L3; Procedure: Herniorrhaphy; Drug: Intravenous (IV) fentanyl; Drug: Bupivacaine
- Five PVB injections (Experimental): Patients will receive five PVB injections between T11 and L3.
  Interventions: Other: Paravertebral block injections between T11 and L3; Procedure: Herniorrhaphy; Drug: Intravenous (IV) fentanyl; Drug: Bupivacaine

INTERVENTIONS:
Other: Paravertebral block injections from T12 to L2 — Three anesthetic injections are done
  Arms: Three PVB injections
Other: Placebo at T11 and L3 — Two injections that contain saline are performed
  Arms: Three PVB injections
Other: Paravertebral block injections between T11 and L3 — Five anesthetic injections are done
  Arms: Five PVB injections
Procedure: Herniorrhaphy — Unilateral inguinal hernia repair
Drug: Intravenous (IV) fentanyl — Patients will be given 1 μg/kg intravenous (IV) fentanyl as premedication
Drug: Bupivacaine — Each patient will receive 75 mg bupivacaine during PVB

SUMMARY:
This prospective double-blinded clinical trial is intended to compare three nerve stimulator- guided paravertebral block injections versus five injections for elderly patients undergoing hernia repair regarding intraoperative hemodynamic stability and postoperative pain.

DETAILED DESCRIPTION:
Introduction

The most effective anesthetic technique for inguinal hernia repair remains a controversial issue; however, paravertebral block (PVB) has resulted in significant postoperative analgesia, less postoperative nausea and vomiting (PONV) and short hospital stay compared to general anesthesia (GA), spinal anesthesia (SA) and ilioinguinal nerve block.

Elderly patients usually have higher risk for developing mental disturbances and cardiopulmonary complications following GA. Hence, elderly patients may benefit from PVB. Although PVB has shown satisfactory outcome; nevertheless, there is no standardized PVB regarding the technique and number of injections.

Based on this background, the objective of this prospective double-blinded study is to compare three nerve stimulator- guided PVB injections versus five injections for elderly patients undergoing hernia repair regarding intraoperative hemodynamic stability and postoperative pain.

Methods Following approval of the Institutional Review Board, written informed consent will be obtained from 200 patients aged above 65 years with ASA II, III or IV admitted to undergo elective unilateral inguinal hernia repair between September 2015 and September 2016.

The sealed envelope technique is used to divide the patients into two groups. Group III (100 patients) will receive three PVB injections from T12 to L2 and placebo at T11 and L3. Group V (100 patients) will receive five PVB injections between T11 and L3. The anesthetist, surgeon, patient and data collector are all blind to the patients' group.

ECG leads, pulse oximetry and non-invasive oscillometric arterial pressure are attached. Patients will be given 1 µg/kg intravenous (IV) fentanyl (Fentanyl Hameln 10 ml, 0.05 mg/ml, Hameln Pharmaceuticals, Germany) as premedication. Unilateral PVB will be performed while the patient is in the lateral decubitus position with the side to be operated being upwards. Sites of injection are marked 2.5-3 cm lateral to the midline of the vertebral column.

Paravertebral block technique Following aseptic preparation of the skin, the injection sites are infiltrated with 0.1 ml of lidocaine 1% each using an 8 mm, 30 G needle (BD Micro-Fine Plus, Becton Dickinson and company, USA). PVB injections are done using a 100 mm 22 G nerve stimulator needle (Stimuplex, B.Braun, Melsungen, Germany). The injections begin at L3 and proceed upwards reaching to T11. The needle is introduced perpendicularly to the skin at the site of the injection point using the following nerve stimulator settings: 5mA, 9V and 2Hz. The stimulating needle is gently manipulated into a position to allow for an adequate muscular response with a stimulating current of 0.4-0.8 mA. Then, the injection is performed. Block onset is determined by cold test and pinprick test.

In order to preserve the double blindness of this clinical trial, two syringes will be used for both groups. The first syringe labeled (A) (20 ml) is filled with 15 mL of solution and used to perform equal injections at the levels T12, L1, and L2 (5mL each). The second syringe labeled (B) (10 ml) is used to inject the solution at the levels T11 and L3 (5 ml each).

To ensure equal anesthetic dose of 75 mg of bupivacaine for each patient, the syringes are prepared as follows:

For group V, both syringes (A) and (B) contain 3mg of bupivacaine/ml whereas for group III, the syringe (A) is prepared with 5 mg bupivacaine/ml while syringe (B) contains placebo.

To allow for adequate blinding, the solution used for injection (saline or local anesthetic mixture) is prepared by an independent nurse outside the operating room.

If a patient feels pain during the surgery, 50 - 100 µg IV fentanyl will be given and followed by 0.4-0.5 mg/kg propofol if needed while keeping the patient responsive to verbal stimulation. If the latter is not sufficient, the patient is converted to GA.

Data Collection Demographic and preoperative variables are collected. Time to perform the block, intraoperative hemodynamic monitoring (MAP and HR) are noted during the entire surgery and recorded pre-incision, at skin incision, at inguinal hernia sac traction, and upon wound closure. Supplemental intraoperative fentanyl and propofol is recorded. Surgery duration, incidence of PONV and numbness are noted.

Patients' satisfaction is also assessed based on their comfort and activity during the procedure, intra- and postoperatively. Patient's comfort is determined by: feeling of pain, PONV, and negative memory of the procedural experience. The patient's activity is based on the ability to sit, move and walk. Patients rate these on a scale of one to three ranging from satisfied, partially satisfied, and unsatisfied. Surgeon's satisfaction is based on the overall intra- and postoperative status of the patient. It is measured based on the following: patient's movement or feeling pain during the operation, self-transportation from the surgical table to stretcher, and postoperative pain.

Postoperative pain is assessed during the first five postoperative days (0 hr, 6 hr, 12 hr, and day 1 till day 5) using the Verbal Numeric Rating Scale (VNRS) (0 no pain and 10 worst possible pain). Patients will be discharged the same day once they had urinated and demonstrated ability to tolerate oral diet. Data will be collected during the hospital stay by residents blind to the patient's group. Patients will be contacted by the same resident during the follow-up period through daily phone calls.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to undergo elective unilateral inguinal hernia repair
* patients with ASA II, III or IV

Exclusion Criteria:

* bilateral inguinal hernia
* incarcerated hernia
* emergency cases
* known history of allergic reactions to local anesthesia
* bleeding disorders
* neurological disorders
* infection at site of injection

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Mean arterial pressure (MAP) for hemodynamic stability | Patients will be monitored during the operation, an expected average of 90 minutes

SECONDARY OUTCOMES:
Pain assessed through the Verbal Numeric Rating Scale (VNRS). | 5 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, Principal Investigator — Chairperson of Anesthesia department
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

REFERENCES:
- [Derived] Naja Z, Kanawati S, Khatib ZE, Ziade F, Nasreddine R, Naja AS. Three versus five lumbar paravertebral injections for inguinal hernia repair in the elderly: a randomized double-blind clinical trial. J Anesth. 2019 Feb;33(1):50-57. doi: 10.1007/s00540-018-2582-9. Epub 2018 Nov 16. PMID 30446826